CLINICAL TRIAL: NCT04737343
Title: The Efficacy of Leflunomide for the Maintenance Therapy of ANCA Associated Vasculitis
Brief Title: Comparison of the Efficacy of Leflunomide and Azathioprine for the Maintenance Therapy of ANCA Associated Vasculitis
Acronym: LEFAZAREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Affiliated Hospital of Jilin University, Changchun,China (Unknown); Second Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Beijing Shijitan Hospital, Capital Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); Sichuan Province People's Hospital (Unknown); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xinping Tian, Professor of Medicine, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR-006
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: ANCA Associated Vasculitis; Maintenance Therapy
Keywords: ANCA Associated Vasculits; Azathioprine; Leflunomide; Maintenance
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Leflunomide; Azathioprine

STUDY DESIGN:
Intervention Model Description: prospective, randomized, open-label, control, non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azathioprine treatment arm (Active Comparator): Patients will be treated with Azathioprine 100mg QD for 18 months combined with rednisone. The dosage of prednisone is tapered in the study period but will be maintained at 7.5mg/d to the end of the study period.All included patients will be treated with TMPco 2 tablets everyday during the study period if not contraindicated or intoleran.t
  Interventions: Drug: Azathioprine Tablets
- Leflunomide treatment arm (Experimental): Patient will be treated with Leflunomide 30mg QD for 18 months combined with prednisone. The dosage of prednisone is tapered in the study period but will be maintained at 7.5mg/d to the end of the study period. All included patients will be treated with TMPco 2 tablets everyday during the study period if not contraindicated or intolerant.
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — Patient will be treated with Leflunomide(Tuoshu, the commericial name) 30mg QD for 18 months
  Other Names: Tuoshu for commericial name
  Arms: Leflunomide treatment arm
Drug: Azathioprine Tablets — Patients included into this study will be treated with Azathioprine tablets 100mg QD for 18 months.
  Arms: Azathioprine treatment arm

SUMMARY:
This study is a prospective, open-labelled, randomized, controlled,multi-center clincial trial. The aim of this study is to verify that the remission rate of patients treated with Leflunomide is not inferior to that of patients treated with Azathioprine.

DETAILED DESCRIPTION:
Background The basic theme of AAV is relapse and remission. The maintenance therapy of AAV aimed to reduce or prevent relapse is very challenge. Although many medications have been used for the maintenance of AAV, Leflunomide (LEF) has not studied thoroughly yet. So far, only one study tested the efficacy of LEF in the maintenance therapy for AAV. However, the sample size of this study is small, so large size clinical study is needed to clarify the role of LEF in the maintenance of AAV.

LEF is one of the most frequently prescribed DMARDs in the treatment of rheumatic diseases in China. It is cheap and widely available. Many experiences have been accumulated about its efficacy and safety in Chinese patients with rheumatic diseases. But there is no study to show its effectiveness in the reduction of the relapse of AAV in China. In this study, we try to compare the effectiveness of LEF and AZA, the gold standard for maintenance therapy, in the maintenance of AAV.

Objectives To verify that the effectiveness of LEF in reducing relapse is not inferior to AZA by comparing the relapse rate of LEF and AZA during the 18 month maintenance treatment of AAV.

Study Design This is a prospective, randomized, open-label, control, non-inferiority study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 to 75 years, both genders can be included.
2. Patients who are newly diagnosed or relapsing granulomatosis with polyangiitis, microscopic polyangiitis, or EGPA in complete remission after combined treatment with glucocorticoids and pulse cyclophosphamide or Rituximab. Remission is defined as a Birmingham Vasculitis Activity Score(BVAS version 3) of 0.
3. Patients must fulfill the 1990 ACR classification criteria of GPA, EGPA and 2012 modified Chapel Hill classification criteria of MPA.
4. Patients have to be ANCA-positive at diagnosis or during the course of their disease.
5. Patients must sign the informed consent.

Exclusion Criteria:

1. Patients with TPMT gene mutation；
2. Patients who had been treated with either AZA or LEF but relapsed in the past;
3. Patients who had been treated with either AZA or LEF but had to stop due to adverse events or intolerance;
4. Patients who have planned for pregnancy in next 2 years;
5. Patients with severe liver dysfunction(defined as the elevation of liver enzyme 3 times the upper limit or Child grade III) or ESRD；
6. Patients with uncontrolled sever hypertension, diabetes, active bacteria or fungal infection;
7. Patients with active hepatitis virus infection as well as patients who have active mycobacteria infection;
8. Patients who are not eligible according to the judge of the principal investigators or site investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients with major relapse in 18 months follow-up time | from inclusion to the end of the study, 18 months in total
  the percentage of patients with major relapse (re-appearance or worsening of disease with a BVAS >0 and involvement of at least one major organ, a life-threatening manifestation, or both) at month 18

SECONDARY OUTCOMES:
The rate of minor relapse of the AZA and LEF treatment group in 18 months. | from inclusion to the end of the study, 18 months in total
  The rate of minor relapse (reappearance or worsening of disease with a BVAS >0, not corresponding to a major relapse but requiring mild treatment intensification) of the AZA and LEF treatment group.
The rate of adverse events and their severity in both LEF and AZA treated patients during 18 months of the study period. | from inclusion to the end of the study, 18 months in total
  2. The rate of adverse events and their severity(Severe events were defined as the adverse events of grade 3 or 4, deaths caused by any cause, cancers, side effects that necessitate hospitalization) in both LEF and AZA treated patients during the study period.
Patients progress to ESRD at the end of the study | from inclusion to the end of the study, 18 months in total
  Patients progress to ESRD at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, Principal Investigator — Peking Unione Mdecial College Hospital
Locations (4):
- China (4):
  - AnHui provincial hospital, Hefei, Anhui
  - the Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - the Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
only patient clincial information coud be released to public